CLINICAL TRIAL: NCT04076384
Title: Effectiveness of a Team-based Follow-up Program in General Practice: Protocol of a Mixed-method Complex Intervention Trial Among People With Chronic Conditions
Brief Title: Effectiveness of a Team-based Follow-up Program in General Practice Among People With Chronic Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bergen University College (Other)
Collaborators: University of Bergen (Other); University of Stavanger (Other)
Responsible Party: Principal Investigator, Beate-Christin Hope Kolltveit, Principal Investigator, Bergen University College
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/28
Record Dates: First submitted 2019-08-26; First posted 2019-09-03 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Type 2; COPD
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pulmonary Disease, Chronic Obstructive | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Team-based consultations (Experimental): Guided Self-Determination
  Interventions: Behavioral: Guided Self-Determination
- Standard care (Experimental): Standard consultation
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Guided Self-Determination — Structured team-based consultations
  Arms: Team-based consultations
Behavioral: Standard care — Standard consultations
  Arms: Standard care

SUMMARY:
The study will develop and evaluate the effectiveness of a team-based follow-up program in general practice (GP) among people with chronic conditions.

DETAILED DESCRIPTION:
The epidemic proportion of lifestyle related non-communicable diseases is a worldwide challenge and public health problem resulting in significant hospitalization rates, mortality and morbidity, and huge personal and societal costs. This project involves research for better public health and health outcomes acknowledging the need for improvements in the health-care services in the prevention of risks and harm and better risk-factor management. We will conduct a randomized control study in four GP practices with ≥3 GPs and ≥one nurse among 154 people at risk for developing Type 2 Diabetes Mellitus (T2DM) or manifest disease, and 154 people in the control group. Inclusion criteria are Diabetes Risc Calculator (FINDRISC) ≥ 15 or HbA1c ≥6,5 % or specific need for individualized follow up such as Body Mass Index (BMI) ≥ 30. In addition, we will conduct a feasibility study among 30 people with risk for Chronic Pulmonary disease (COPD) or manifest disease. The study has the following two objectives: 1) to evaluate the effectiveness of a team-based follow-up program among people with risk for T2DM or manifest T2DM with the use of Guided Self-Determination (GSD) as an empowerment approach for patients in general practice, 2) to test the feasibility and pilot a team-based follow-up program among people with risk for COPD or manifest COPD with the use of GSD as an empowerment approach for patients in general practice.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20-80 years with FINDRISC score ≥15
* Body Mass Index ≥ 30
* Manifest T2DM (HbA1c ≥48 mmol/mol (6,5%))
* Positive smoking status (risk for COPD)
* Manifest COPD (spirometry value: FEV1/FVC < 0,7).

Exclusion Criteria:

* Severe somatic disease (cancer, end stage renal disease)
* Severe psychiatric diagnosis or dementia
* Patients who do not understand nor speak Norwegian.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Patient Activation Measure (PAM-13) | 12 months
  The Patient Activation Measure instrument capture patient's knowledge, skills and confidence for self-management living with chronic conditions.It has four response categories with scores from 1 to 4: "strongly disagree" (1), "disagree" (2), "agree" (3) and "agree strongly" (4). The scale scores are transformed to a 0 to 100 scale (0 = lowest activation level, 100 = highest activation level).

SECONDARY OUTCOMES:
HbA1c | 12 months
  Blood glucose
Problem Areas in Diabetes Scale (PAID-5) | 12 months
  The Problem Areas in Diabetes Scale measures negative emotions related to living with diabetes. The scores are on a 5-point Likert scale ranging from 0 (not a problem) to 4 (a serious problem). Scale scores are transformed to a 0-100 scale, with higher scores indicating greater emotional problems.
The World Health Organization 5-item Well-Being Index (WHO-5) | 12 months
  The World Health Organization 5-item Well-Being Index (WHO-5) measures subjective psychological well-being by means of five positively worded items reported on a 6-point Likert scale ranging from 0 (not present) to 5 (constantly present). An overall score is calculated as the sum of the five items and rescaled to values ranging from 0 to 100. Higher scores represent better emotional well-being.
Quality of Life-BREF 2-Item questionnaire | 12 months
  The WHO Quality of Life-BREF questionnaire comprises two items indicating better overall quality of life or general health. Both are rated on a 5-point Likert scale with higher scores indicating better overall quality of life or general health.
The EuroQol EQ-5D-5L | 12 months
  The EuroQol EQ-5D-5L consists of five item dimensions measuring general health. Ratings are on a Likert scale from 1-5 with higher scores indicating more difficulties. The EQ-5D also comprises a visual analogue scale from 1 (worst possible health) to 100 (best possible health).
The European Health Literacy survey tool (HLS-EU-Q12) | 12 months
  The European health literacy survey tool measures people's knowledge, motivation and competences to access, understand, appraise, and apply health information.The ratings are on a four-point rating scale, with response categories from 1 (very easy) - 4 (very difficult). Higher scores indicate lower health literacy.
Perceived Competence for Diabetes Scale (PCDS) | 12 months
  The Perceived Competence for Diabetes Scale (PCDS) contains four items and assesses the degree of competence perceived by persons with diabetes to manage the daily aspects of diabetes care. The scores are on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Higher scores represent greater perceived competence.
The Finnish Diabetes Risc Calculator (FINDRISC) | 12 months
  The Finnish Diabetes Risc Calculator identify people at increased risk for future type 2 diabetes The different items are weighted into a total score ranging from 0 to 26 points with higher scores indicating greater individual 10-year risk of developing type 2 diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Beate-Christin H Kolltveit, Ph.D, Principal Investigator — Western Norway University of Applied Sciences
Locations (1):
- Western Norway University of Applied Sciences, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kolltveit BH, Oftedal BF, Thorne S, Lomborg K, Graue M. Experiences of an interprofessional follow-up program in primary care practice. BMC Health Serv Res. 2024 Feb 23;24(1):238. doi: 10.1186/s12913-024-10706-9. PMID 38395910
- [Derived] Kolltveit BH, Graue M, Borge CR, Frisk B. Patients' experiences with participating in a team-based person-centred intervention for patients at risk of or diagnosed with COPD in general practice. Pilot Feasibility Stud. 2023 Sep 25;9(1):164. doi: 10.1186/s40814-023-01398-9. PMID 37749601